CLINICAL TRIAL: NCT04942847
Title: Application of Cognitive Combined Sucking Task Training in Dysphagia After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-721
Record Dates: First submitted 2021-05-29; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-05

CONDITIONS: Prospective Study

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (No Intervention): The control group received routine nursing, including diet nursing, life nursing, direct and indirect training, health education and so on. Patients were followed up regularly by telephone after discharge
- Dual task training group (Experimental): On the basis of routine swallowing function training, the use of sucking training rehabilitation device is mainly used for tongue muscle training and lip muscle training to improve the control and delivery ability of tongue muscle to food.At the same time,adopt Troup's playing and comprehensive analysis ability training.Disrupt the three sets of cards, instruct the patient to read words or say colors, and measure the patient's reaction time with an electronic timer.Comprehensive analysis ability training: including digital training or item classification training.
  Interventions: Device: Sucking trainer; Device: Cognitive card

INTERVENTIONS:
Device: Sucking trainer — Repeated sucking for tongue flexibility training can improve the tongue muscle's ability to control and transmit food, and improve the swallowing function.
  Arms: Dual task training group
Device: Cognitive card — To measure the patient's ability to focus, to calculate, to remember and to judge
  Arms: Dual task training group

SUMMARY:
this topic research, on the basis of traditional swallowing training to develop a set of scientific and advanced type of swallowing disorder in patients with stroke rehabilitation training of the new strategy, combined with cognitive training and sucking training for swallowing disorder in patients with cerebral apoplexy and to provide professional, systematic and comprehensive rehabilitation guidance, promote patients early recovery and return to society.

DETAILED DESCRIPTION:
The incidence of dysphagia in stroke patients is as high as 30% ~ 65%. Dysphagia caused by stroke is the primary cause of dysphagia and an independent risk factor for the prognosis of patients. The rehabilitation of cognitive function is the key to the assessment of swallowing and the recovery of rehabilitation function after stroke, and complete consciousness, sensorimotor consciousness and motivation are the prerequisites for the rehabilitation of swallowing function. Traditional rehabilitation programs focus more on the single task training of patients' function and ignore the training of cognitive function. Cognitive deglutition dual task training is a kind of cognitive rehabilitation training at the same time of deglutition rehabilitation treatment. In this study, the "dual task" training mode of cognitive combined sucking training was applied to the rehabilitation of patients with swallowing dysfunction after stroke, to evaluate the rehabilitation of patients with swallowing function and cognitive function, and to further guide the clinical development and implementation of early rehabilitation treatment and nursing.

Expected results:

Through this topic research, on the basis of traditional swallowing training to develop a set of scientific and advanced type of swallowing disorder in patients with stroke rehabilitation training of the new strategy, combined with cognitive training and sucking training for swallowing disorder in patients with cerebral apoplexy and to provide professional, systematic and comprehensive rehabilitation guidance, promote patients early recovery and return to society.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Acute stroke
* Clinical diagnosis of Deglutition disorders
* Must be able to communicate through reading and writing

Exclusion Criteria:

* Dysphagia not caused by stroke Patients
* With important organ failure or critical illness
* Severe mental illness or cognitive impairment
* Severe oropharyngeal organic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cognitive function at 7 days | Within 8 hours after admission and 7 days after admission
  MMSE(Mini-mental State Examination) score, composed of 20 questions, can be used to evaluate orientation, attention, calculation ability, long-term and short-term memory and judgment ability. The score ranges from 0 to 30, The lower the score, the more serious the cognitive impairment.
Change from Baseline Swallowing function at 7 days | Within 8 hours after admission and 7 days after admission
  (Swallowing-Quality of Life)SWALQO score. has 44 items, which are used to evaluate 11 aspects of quality of life of patients with dysphagia.the total score was converted into 0-100. 0 means that the quality of life is extremely low, 100 means that the quality of life is normal, and the higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Qiaomin Tang, Principal Investigator — 2nd Affiliated Hospital,School of Medicine,Zhejiang University,China
Locations (1):
- 2nd Affiliated Hospital,School of Medicine,Zhejiang University,China, Hangzhou, Zhejaing, China

IPD SHARING:
Plan to Share IPD: Yes